CLINICAL TRIAL: NCT03939429
Title: A Phase 1, Randomized, Double-Blind, Placebo-Controlled, Ascending Single and Multiple-Dose Study of the Safety, Tolerability, Pharmacokinetics of Oral QPX2015 in Healthy Adult Subjects
Brief Title: Phase 1 Study of Oral QPX2015 in Healthy Adult Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Qpex Biopharma, Inc. (Industry)
Collaborators: Biomedical Advanced Research and Development Authority (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Qpex-100
Record Dates: First submitted 2019-05-01; First posted 2019-05-06 (Actual); Last update posted 2022-10-10 (Actual); Status verified 2019-05

CONDITIONS: Bacterial Infections
Keywords: beta-lactam antibiotic
MeSH Terms: conditions — Bacterial Infections | interventions — Contraceptives, Oral

STUDY DESIGN:
Intervention Model Description: double-blind, placebo controlled ascending single- and multiple-dose
Who Masked: Participant, Investigator
Masking Description: double-blind, placebo controlled ascending single- and multiple-dose
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- QPX2015 (Experimental): QPX2015, antibiotic
  Interventions: Drug: QPX2015
- Placebo (Placebo Comparator): Matched placebo
  Interventions: Drug: Placebo oral capsule

INTERVENTIONS:
Drug: QPX2015 — antibiotic
  Other Names: oral dose
  Arms: QPX2015
Drug: Placebo oral capsule — Placebo comparator
  Other Names: oral dose
  Arms: Placebo

SUMMARY:
QPX2015 (beta-lactam antibiotic) is being studied at higher than approved doses to combine with a new beta-lactamase inhibitor to treat bacterial infections, including those due to multi-drug resistant bacteria.

DETAILED DESCRIPTION:
The worldwide spread of resistance to antibiotics among gram-negative bacteria, particularly members of the ESKAPE group of pathogens, has resulted in a crisis in the treatment of both hospital acquired and community acquired infections. In particular, the increase in Enterobacteriaceae expressing extended spectrum beta-lactamases (ESBLs) and carbapenemases that are resistant to all oral beta-lactams and fluoroquinolones in the community have resulted in many patients requiring admission just for IV antibiotics to treat their infections.

Qpex Biopharma is developing a fixed combination antibiotic of QPX2015 (beta-lactam antibiotic) plus a new beta-lactamase inhibitor.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy adult males and/or females of non-child bearing potential, 18 to 55 years of age (inclusive).
2. Body mass index (BMI) ≥ 18.5 and ≤ 29.9 (kg/m2) and weight between 55.0 and 100.0 kg (inclusive).
3. Medically healthy with clinically insignificant screening results (e.g., laboratory profiles, medical histories, electrocardiograms [ECGs], physical examination) as assessed by the PI.
4. Voluntarily consent to participate in the study.
5. If male, agree to be sexually abstinent or agree to use two approved methods of contraception when engaging in sexual activity from study check-in through completion of the end-of-study. Subjects must agree to use two approved methods of contraception for 30 days following the last administration of the study drug, and to not donate sperm during this same period of time. In the event that the sexual partner is surgically sterile, contraception is not necessary.
6. Females of non-childbearing potential with serum FSH levels ≥ 40 mIU/mL are either postmenopausal (defined as 12 months spontaneous amenorrhea) or have undergone sterilization procedures at least 6 months prior to dosing.

Exclusion Criteria:

1. History or presence of significant cardiovascular, pulmonary, hepatic, renal, hematological, gastrointestinal, endocrine, immunologic, dermatologic, neurological, or psychiatric disease.
2. Positive urine drug/alcohol testing at screening or check-in (Day -1).
3. Positive testing for HIV, hepatitis B or C
4. History or presence of alcoholism or drug abuse within last 2 years
5. Use of more than 5 packs/week of tobacco/nicotine-containing product within last 6 months prior dosing.
6. Use of any prescription medication (with the exception of hormonal contraceptives or hormone replacement therapy for females) within 14 days prior to dosing.
7. Use of any over-the-counter (OTC) medication, including herbal products and vitamins, within the 7 days prior to dosing.
8. Use of antacids, H2 receptor blockers or proton pump inhibitors 3 days prior to dosing.
9. History of any hypersensitivity or allergic reaction to cephalosporins, penicillins, carbapenems, or monobactams).
10. Participation in another investigational clinical trial within 30 days prior to Dosing or within 5 half-lives of the previous investigational drug, whichever is longer.
11. Females who are pregnant or lactating.
12. QTcF interval >450 msec, or history of prolonged QT syndrome at screening or check-in
13. Calculated creatinine clearance less than 80 mL/min (Cockcroft-Gault method) at screening or check-in.
14. Subjects who have any clinically significant abnormalities on laboratory values: White blood cell count < 3,000/mm3, hemoglobin < 11g/dL or Absolute neutrophil count < 1,200/mm3 or platelet count < 120,000/mm3.
15. Liver function abnormalities defined by an elevation in bilirubin, AST or ALT 1.5 x ULN of the normal range for subjects based on age and sex.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2019-05-20 (Actual); Primary Completion 2019-10-06 (Actual); Study Completion 2019-10-06 (Actual)

PRIMARY OUTCOMES:
Incidence of Treatment -Emergent Adverse events by subject and by cohort | Study Day 1 to 13
  Number of patients with Treatment-Emergent AEs by treatment arm, severity and relationship to treatment
Number of patients with changes from baseline in safety parameters | Study Day 1 to 13
  Number of patients with changes in safety parameters before and after dosing by subject and treatment arm
Peak plasma Concentration measurements by subject and by cohort (Cmax) | Study Day 1 to 13
  Comparison will be performed between the cohorts for Cmax. Mean graphical presentation of the data will be reported. Statistical analysis of exposure parameters will be performed.
Time concentration data measurements by subject and by cohort (Tmax) | Study Day 1 to 13
  Comparison will be performed between the cohorts for Tmax.
Area under the plasma concentration versus time curve (AUC) between cohorts | Study Day 1 to 13
  Comparison will be performed between the cohorts for AUC. Mean graphical presentation of the data will be reported. Statistical analysis of exposure parameters will be performed.
Urine PK amount excreted by subject and by cohort | Study Day 1 to 13
  Urine PK parameters such as amount excreted will be calculated from urinary excretion data
Urine PK % dose excreted by subject and by cohort | Study Day 1 to 13
  Urine PK parameters such as amount of % dose excreted will be calculated from urinary excretion data

CONTACTS AND LOCATIONS:
Overall Officials: Jeffery S Loutit, MBChB, Study Director — Qpex Biopharma, Inc.
Locations (1):
- CMAX, Adelaide, South Australia, Australia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Hernandez-Mitre MP, Wallis SC, Morgan EE, Dudley MN, Loutit JS, Griffith DC, Roberts JA. A phase I, randomized, double-blind, placebo-controlled, ascending single- and multiple-dose study of the pharmacokinetics, safety, and tolerability of oral ceftibuten in healthy adult subjects. Antimicrob Agents Chemother. 2024 Jan 10;68(1):e0109923. doi: 10.1128/aac.01099-23. Epub 2023 Dec 7. PMID 38059635